CLINICAL TRIAL: NCT03080467
Title: Long-term Outcome of the Primary Wound Repair of Traumatic Skin Lacerations in the Head Area in Pediatric Patients: Suture Versus Tissue Adhesive
Brief Title: Long-Term Outcome of Pediatric Traumatic Wound Repair: Suture Versus Tissue Adhesive
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-01304
Record Dates: First submitted 2017-03-09; First posted 2017-03-15 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Tissue Adhesives; Laceration; Sutures; Wounds and Injuries; Child
Keywords: Trauma; Laceration; Suture; Cosmesis; Ethyl-2-Cyanoacrylate; Tissue adhesive; Lip lacerations; Skalp lacerations; Facial injuries
MeSH Terms: conditions — Lacerations; Wounds and Injuries; Facial Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Suture: Wound repair with suture
- Tissue adhesive: Wound repair with tissue adhesive

SUMMARY:
This project is an observational trial investigating wound cosmetic appearance after repair of traumatic skin lacerations in the head area of pediatric patients with two different approaches to skin closure: sutures versus tissue adhesive. Photographs will be taken at two follow-up visits after repair and later assessed by external blinded plastic surgeon using standard cosmetic assessment scales. The investigators hypothesize that cosmetic wound outcome will be equivalent in these two wound repair treatment options.

DETAILED DESCRIPTION:
Investigation of the long-term outcome of 300 pediatric patients with traumatic skin lacerations in the head area. After primary wound repair with suture or with tissue adhesive, eligible patients will be enrolled on the emergency department (baseline visit). The second follow-up visit will take place 5-10 days after the baseline visit and the third follow-up visit will be completed 6-12 months after trauma. At both follow-up visits, clinical examination and a brief interview will be performed. Photo documentation is completed at both the baseline and the follow-up visit.

Encrypted photo documentation will be evaluated by blinded external plastic surgeons. Primary Outcome is the cosmetic appearance using standard assessment scales, secondary outcomes are the occurrence of complications, cost-effectiveness and patient's satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* 0 till16 years of age
* Any primary wound repair treatment of a laceration caused by trauma and involving the skin of the head area
* Patient or caregiver must be able to understand and sign an informed consent

Exclusion Criteria:

* Pre-existing conditions that affect wound healing adversely
* Patients who demonstrate severe or life-threatening injuries
* Patients / caregivers with communication / logistic barriers that would make them unfit to provide informed consent or to attend the follow-up visits

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients after completion of a primary wound repair treatment with suture or tissue adhesive in the Pediatric Emergency Unit
Sampling Method: Non-Probability Sample
Enrollment: 386 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Cosmetic scar appearance | second follow-up visit: 6 till 12 months after wound repair
  Cosmetic appearance will be assessed using the modified Patient and Observer Scar Measurement Score

CONTACTS AND LOCATIONS:
Overall Officials: Clemens M Schiestl, PD, Principal Investigator — Children's University Hospital of Zurich
Locations (1):
- Children's University Hospital of Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Farion K, Osmond MH, Hartling L, Russell K, Klassen T, Crumley E, Wiebe N. Tissue adhesives for traumatic lacerations in children and adults. Cochrane Database Syst Rev. 2002;2002(3):CD003326. doi: 10.1002/14651858.CD003326. PMID 12137689
- [Background] Singer AJ, Hollander JE, Quinn JV. Evaluation and management of traumatic lacerations. N Engl J Med. 1997 Oct 16;337(16):1142-8. doi: 10.1056/NEJM199710163371607. No abstract available. PMID 9329936
- [Background] Idriss N, Maibach HI. Scar assessment scales: a dermatologic overview. Skin Res Technol. 2009 Feb;15(1):1-5. doi: 10.1111/j.1600-0846.2008.00327.x. PMID 19152571
- [Background] Fearmonti R, Bond J, Erdmann D, Levinson H. A review of scar scales and scar measuring devices. Eplasty. 2010 Jun 21;10:e43. PMID 20596233
- [Background] Fearmonti RM, Bond JE, Erdmann D, Levin LS, Pizzo SV, Levinson H. The modified Patient and Observer Scar Assessment Scale: a novel approach to defining pathologic and nonpathologic scarring. Plast Reconstr Surg. 2011 Jan;127(1):242-247. doi: 10.1097/PRS.0b013e3181f959e8. PMID 21200219
- [Background] Brown BC, Moss TP, McGrouther DA, Bayat A. Skin scar preconceptions must be challenged: importance of self-perception in skin scarring. J Plast Reconstr Aesthet Surg. 2010 Jun;63(6):1022-9. doi: 10.1016/j.bjps.2009.03.019. Epub 2009 Jun 5. PMID 19501559
- [Background] Lewis-Jones MS, Finlay AY. The Children's Dermatology Life Quality Index (CDLQI): initial validation and practical use. Br J Dermatol. 1995 Jun;132(6):942-9. doi: 10.1111/j.1365-2133.1995.tb16953.x. PMID 7662573
- [Background] Olsen JR, Gallacher J, Finlay AY, Piguet V, Francis NA. Quality of life impact of childhood skin conditions measured using the Children's Dermatology Life Quality Index (CDLQI): a meta-analysis. Br J Dermatol. 2016 Apr;174(4):853-61. doi: 10.1111/bjd.14361. Epub 2016 Mar 6. PMID 26686685
- [Derived] Fontana S, Schiestl CM, Landolt MA, Staubli G, von Salis S, Neuhaus K, Mohr C, Elrod J. A Prospective Controlled Study on Long-Term Outcomes of Facial Lacerations in Children. Front Pediatr. 2021 Feb 12;8:616151. doi: 10.3389/fped.2020.616151. eCollection 2020. PMID 33643965